CLINICAL TRIAL: NCT05975177
Title: Evaluation of the Efficacy and Safety of STERIFY GEL in the Treatment of Periodontitis Following Scaling and Root Planing: Pivotal, Prospective, Single-center, Split-mouth, Randomized, Controlled Study
Brief Title: Evaluation of the Efficacy of STERIFY GEL in the Treatment of Periodontitis Following Scaling and Root Planing
Acronym: SFYCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sterify S.r.l. (Industry)
Collaborators: Sciently di Omar Sabry (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFYCT
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Parodontitis
Keywords: Sterify gel; periodontal disease; periodontal pockets; scaling and root planing; oral health; dental care
MeSH Terms: conditions — Dry Socket; Periodontal Diseases; Periodontal Pocket | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: The study is a split-mouth study. STERIFY GEL will be administered into the periodontal pockets of one or two segments of patients undergoing whole-mouth extended SRP, with the contralateral segments serving as controls (split-mouth), in a single session.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sterify Gel + SRP (Experimental): Scaling and root planing in the assigned site, followed by intra-pocket administration of Sterify Gel, applied to the bottom of the pocket until the gel emerges or becomes visible at the gingival margin
  Interventions: Device: Sterify Gel; Procedure: Scaling and root planing
- SRP only (Active Comparator): Scaling and root planing in the assigned site.
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Device: Sterify Gel — A mucoadhesive polymeric hydrogel in a prefilled syringe for nonsurgical treatment of periodontal and peri-implant pockets, composed of polyvinyl polymers, hydroxytyrosol, nisin, and magnesium ascorbyl phosphate
  Arms: Sterify Gel + SRP
Procedure: Scaling and root planing — The non-surgical procedure involved SRP under local anesthesia with EMS scalers and Gracey curettes.

SUMMARY:
The purpose of this clinical study is to evaluate the safety and efficacy of treating periodontal disease with the STERIFY GEL medical device in combination with SRP procedure, in terms of periodontal pocket healing. Efficacy will be compared with the use of the nonsurgical SRP technique alone, which is considered a gold standard treatment for periodontitis, with the aim of observing improved results when using the STERIFY GEL device.

The study is prospective, split-mouth.STERIFY GEL will be administered into the periodontal pockets of one or two segments of patients undergoing whole-mouth extended SRP, with the contralateral segments serving as controls (split-mouth), in a single session.

DETAILED DESCRIPTION:
The purpose of the study is to test the safety and efficacy of STERIFY GEL in promoting healing of periodontal pockets following SRP, compared with treatment with SRP alone. With specific visco-elastic and mucoadhesive properties, STERIFY GEL easily penetrates into the deepest and hard-to-reach areas of periodontal and peri-implant pockets, adhering to the gingival tissue and alveolar bone, providing complete coverage of the pockets. The effect of STERIFY GEL is promoted by a physical mechanism of action. After SRP, the gel is applied into the gingival pocket, where it acts primarily as a filler to restore volume, physically preventing bacteria from entering and reinfecting the pocket. STERIFY GEL can thus mechanically protect treated pockets and bone defects, promoting tissue healing. The occluding action at the level of periodontal and peri-implant gingival pockets, in synergy with the accessory action of hydroxytyrosol, nisin, and magnesium ascorbyl phosphate, prevents bacterial recolonization and promotes subsequent tissue regeneration.

Although SRP surgery is considered a gold standard treatment for periodontitis, it may in some cases be insufficient to decontaminate the pocket allowing bacteria to recolonize the tissues promoting new inflammation that can worsen the clinical picture.STERIFY GEL may find useful application in cases of moderate to severe chronic periodontal disease as an adjunctive treatment following SRP to improve and accelerate healing parameters and prevent recurrent inflammation and infection.In addition, antimicrobial control action prevents antibiotic use and the risk associated with antibiotic resistance.Such control of periodontal disease also allows for the maintenance of patients who cannot undergo surgical treatment (e.g., patients on bisphosphonate therapy, defected etc.).

ELIGIBILITY:
Inclusion Criteria:

* Patients with grade III and IV chronic periodontal disease according to the European Federation of Periodontology classification involving at least two sites
* Adherence to the study and signing of informed consent
* Major age- Participants with a minimum of 6 teeth with periodontal pocket depth greater than 5mm- Participants with at least 20 teeth

Exclusion Criteria:

* Established hypersensitivity to one or more components of the device- Pregnancy or lactation- Heavy smoker (more than 9 cigarettes per day)- Concomitant dental disease, except periodontitis, or planned treatment that may interfere with the study or study procedure, such as dental surgery or tooth implantation- Diabetes mellitus, rheumatoid arthritis, or other chronic diseases that may affect disease or treatment
* Aggressive periodontitis
* History of radiation or chemotherapy
* Autoimmune mucosal diseases
* Mental illnesses
* Parafunctions such as bruxism
* Use of antibiotics in the past 3 months
* Periodontal surgeries in the past 12 months in the areas covered by the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-12-03 (Actual); Primary Completion 2023-03-11 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Pocket Depth | Pre-treatment, 1 month, 2 months, 3 months
  Measurement by periodontal probe of periodontal pocket depth. Unit of measurement in mm with a sensitivity of 0.5 mm.

SECONDARY OUTCOMES:
Gingival recession | Pre-treatment, 1 month, 2 months, 3 months
  Measurement by periodontal probe of the distance from the cemento-enamel junction to the depth of the free gingival margin.
Clinical Attachment Level | Pre-treatment, 1 month, 2 months, 3 months
  Measurement by periodontal probe of the distance in millimeters between the amelo-cement junction (the boundary between the crown and root of the tooth) and the bottom of the pocket.It can also be calculated by summing the gingival recession and the periodontal pocket.
Plaque Index | Pre-treatment, 1 month, 2 months, 3 months
  The plaque index (PI) (Silness J & Löe H), is recorded, during the clinical periodontal examination, at 4 to 6 sites for each tooth element present by circumferential probing with a manual periodontal probe.The 6 dental sites considered are: buccal, mesio-buccal, disto-buccal, lingual, mesio-lingual, and disto-lingual (if there are 4: distal, proximal, palatine/lingual, buccal).Each site is given a score from 0 to 3, where: 0 no plaque, 3 abundance of plaque.
Bleeding Index | Pre-treatment, 1 month, 2 months, 3 months
  % measurement. Each site is gently probed with a periodontal probe at six sites (mesial, middle, and distal on both buccal and lingual surfaces): bleeding is assessed as present or absent, and the number of sites where bleeding is present is recorded.The number of sites where bleeding is recorded is divided by the total number of sites available in the mouth and multiplied by 100 to express the bleeding index as a percentage.
Furcations | Pre-treatment, 1 month, 2 months, 3 months
  0: no furcation1: horizontal loss of supporting tissues not exceeding one third of the tooth width 2: horizontal loss of supporting tissues exceeding one-third of the tooth width but not affecting the entire furcation 3: Horizontal loss of supporting tissues "passing through" the entire furcation area.
Grade of Mobility | Pre-treatment, 1 month, 2 months, 3 months
  The survey of dental mobility completes the objective examination. It is important to remember that mobility can be periodontal, traumatic, or endodontic in origin and should be assessed by the application of slight forces conveyed through two instruments and not with the fingers.
  Class 0: physiological mobility.Class 1: slightly increased mobility, slight horizontal displacements (Perceptible mobility <1mm in buccolingual direction) Class 2: markedly increased mobility without functional impediment, displacements in horizontal direction (>1mm but <2mm) Class 3: markedly increased mobility with functional impediment, displacements even in vertical direction (>2mm or depressibility in the socket)
Quantification of bacterial contamination | Pre-treatment, 3 months
  Bacterial contamination assessed through quantitative PCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Odontostomatologia, ASST dei Sette Laghi, Varese, Italy

IPD SHARING:
Plan to Share IPD: No